CLINICAL TRIAL: NCT03370614
Title: Pilot Study of the Physiological Effects of an Integrative Medicine Approach in Irritable Bowel Syndrome
Acronym: IBS
Status: Active, not recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 17D.184
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: PET; MRI; Irritable Bowel Syndrome; Irritable Bowel; Positron emission tomography; Magnetic resonance imaging; FDG; Fluorodeoxyglucose
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS Group: Participants will complete initial baseline and follow up IBS evaluations and questionnaires. Pre and Post FDG-PET-MR scans will be conducted to evaluate changes at baseline and approximately 2 months after dietary and nutritional counseling.
  Interventions: Other: IBS Group
- Healthy Control Group: Participants will complete initial baseline evaluations and questionnaires. Participants will also receive a FDG-PET-MR scan.
  Interventions: Other: Healthy Control Group

INTERVENTIONS:
Other: IBS Group — Participants will receive approximately 2 months of dietary and nutritional counseling.
  Groups: IBS Group
Other: Healthy Control Group — Participants will not receive any dietary or nutritional counseling.
  Groups: Healthy Control Group

SUMMARY:
Although underutilized, what is emerging as one of the best ways of evaluating inflammation in the body, particularly in difficult to observe regions, is through the use of Fluorodeoxyglucose (FDG) positron emission tomography (PET). FDG is taken up in the body much like glucose and is particularly taken up in areas of inflammation where there is increased metabolism. Therefore, this technology can be used to assess inflammation, and measure the reduction in inflammation as the result of integrative interventions that target dietary modifications designed to reduce inflammation. With this proposed study, we plan to use FDG PET-MRI technology to develop a more specific and sensitive approach for evaluating areas of inflammation associated with IBS and measuring improvements in that inflammation in response to effective integrative interventions.

DETAILED DESCRIPTION:
The typical goal of the integrative medicine approach is to develop an individualized plan to help restore homeostasis to the gastrointestinal system targeting a reduction in inflammation as an important element in helping to relieve symptoms. One of the most problematic issues though is to determine where in the GI tract the inflammation is occurring and then evaluating improvements in inflammation as any intervention proceeds.

Participants will undergo a small battery of diagnostic tests that include magnetic resonance imaging (MRI), fluorodeoxyglucose positron emission tomography (FDG-PET). A secondary goal of this study is to evaluate the utility of FDG PET-MRI for assessing reductions in inflammation in patients managed with an integrative medicine approach based upon diet and nutritional counselling.

ELIGIBILITY:
Inclusion Criteria for IBS Subjects:

1. Age greater than 18 years old.
2. Meets the Rome III criteria for IBS: Recurrent abdominal pain or discomfort at least 3 days per month in the last 3 months associated with 2 or more of the following: 1) Improvement with defecation; 2) Onset associated with a change in frequency of stool; 3) Onset associated with a change in form (appearance) of stool.
3. Patients have no other pre-existing and active significant gastrointestinal medical, neurological, or psychological disorders as per review by the PI
4. Minor, stable health problems that should have no substantial effect on cerebral blood flow will be allowed (i.e. controlled hypertension, medication controlled diabetes) as per review by the PI.
5. Patients will be allowed to be taking medications or supplements at the initial intake, but they must be on a stable dose regimen for at least 1 month.
6. Able to give informed consent and willing to complete the study.

Inclusion criteria for Healthy Controls:

1. No significant current active medical conditions.
2. Stable medical conditions as determined by the PI are allowed.
3. No brain or body abnormalities that would affect the acquisition or analysis of the scan.

Exclusion Criteria for IBS Subjects and Healthy Controls:

1. Previous abdominal (bowel) surgery.
2. Not continuously taking antioxidants or anti-inflammatory medications ( to be reviewed by the PI.
3. No other active medical conditions potentially requiring changes in treatment regimen during the study duration.
4. Not pregnant or breast feeding
5. Enrollment in active clinical trial/ experimental therapy within the prior 30 days.
6. Subject is unable or unwilling to lie still in the scanner (i.e. due to claustrophobia or weight > 350 pounds)
7. Subject has metal in their body or other reason that they cannot undergo magnetic resonance imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited only if they experience symptoms of IBS.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Combined PET/MRI to define IBS activity and inflammation pattern. | Baseline and 2 months
  To use PET-MRI to define abnormal brain and body activity and evaluate changes in inflammation for IBS patients.

SECONDARY OUTCOMES:
Use combined PET/MRI to demonstrate brain and body activity in responders and non-responders. | Baseline and 2 months
  Patterns will be compared between those who respond and those who do not respond to dietary/nutritional program.

OTHER OUTCOMES:
Beck Depression Inventory. | Baseline and 2 months
  This assessment questionnaire will be used as one of the evaluation questionnaires for the study.
Standard Form (SF) 36 | Baseline and 2 months
  This 36 item assessment questionnaire will be used as one of the evaluation questionnaires for the study.
Profile of Mood Scale | Baseline and 2 months
  The Profile of Mood States (POMS) is a questionnaire of 65 single word items that asks "How have you been feeling in the past week including today." The subjects will select their response to each word that describes a mood or feeling on a Lickert scale from 1= Not at All, 2= A Little, 3=Moderately, 4=Quite a lot, to 5=Extremely. The responses are scored to generate values for Tension, Anger, Confusion, Depression and Vigor. The higher scores indicate a greater presence of that mood or state.
Self-Evaluation Questionnaire | Baseline and 2 months
  This assessment questionnaire will be used as one of the evaluation questionnaires for the study.
Symptom Diary | Baseline and 2 months
  This assessment questionnaire will be used as one of the evaluation questionnaires for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B. Newberg, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Villanova, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03370614/ICF_003.pdf